CLINICAL TRIAL: NCT01115413
Title: Influence of Young Maternal Age on Pregnancy Outcome in Central Europe
Brief Title: The Effect of Teenage Maternity on Obstetrical and Perinatal Outcomes
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Daniel Alexander Beyer, Dr. D. A. Beyer, University of Luebeck
Other Study IDs: UKSH-HL-10-064
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy
Keywords: teenage; pregnancy; obstetrical risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- young maternal age: maternal age of < 18 years
- adult maternal age: maternal age >/= 18 years

SUMMARY:
The purpose of this study is to estimate the effect of maternal teenage on pregnancy and perinatal outcomes among Caucasian pregnant women.

DETAILED DESCRIPTION:
During the past decade in the United States, approximately 10 percent of teenage girls from 15 to 19 became pregnant. According to the National Vital Statistics Report 2009 seventy of one thousand births in the United States accounted to teenagers from 15 to nineteen years of age during in 2005 and fell to forty per 1,000 women in 2006. In contrary, the overall teenage birth rate lay at twenty- two per 1,000 births in Massachusetts in 2007 ranging from seventy to thirteen per 1,000 women for Hispanic vs. white women aged 15- 19 years. Central European data showed equal results for teenage pregnancy birth rates. According to the German National Institute of Vital Statistics thirty-four of one thousand births in Germany accounted to teenagers younger than 20 years of age. This pattern is a source of concern since teenage mothers have an increased risk of having low-birth- weight babies, premature babies, and babies who die during the first year of life. Additionally, teenage mothers are more likely to suffer from other concomitant pregnancy diseases such as preeclampsia or anemia.

Furthermore, teenage mothers are more likely than older mothers to be poor, less well educated, non- white, unmarried and they are less likely to have received early prenatal care. Dealing with pregnant adolescents therefore means a great challenge in modern obstetrics. Previous research has shown racial differences as well as weight differences for increased risk of adverse prenatal outcome among African Americans and teenagers. Taking into account the impact of race on pregnancy outcomes, our goal was to examine the relationship of young maternal age on obstetrical outcomes in a predominantly Caucasian central European teenaged population.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity
* Maternal age of < 18 years for group A and
* Maternal age >/= 18 years for group B

Exclusion Criteria:

* Preterm delivery < 24 + 0 weeks of gestation post menstruation
* Confirmed multiple pregnancy
* Maternal and fetal co morbidity
* Presentation other than cephalic presentation and incomplete data

Ages: 11 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: retrospective cohort analysis of all deliveries at the Schleswig-Holstein University Hospital Center in Lübeck from January 2000 through December 2009
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
mode of delivery | 9yrs

SECONDARY OUTCOMES:
time of labor | 9yrs
maternal injury during labor and delivery | 9yrs
neonatal outcome | 9yrs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Beyer, M.D., Principal Investigator — Lübeck University
Locations (1):
- Schleswig- Holstein University, Campus Lübeck, Department of Obstetrics and Gynecology, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Picklesimer AH, Jared HL, Moss K, Offenbacher S, Beck JD, Boggess KA. Racial differences in C-reactive protein levels during normal pregnancy. Am J Obstet Gynecol. 2008 Nov;199(5):523.e1-6. doi: 10.1016/j.ajog.2008.04.017. Epub 2008 Jun 9. PMID 18539258
- [Background] Steinfeld JD, Valentine S, Lerer T, Ingardia CJ, Wax JR, Curry SL. Obesity-related complications of pregnancy vary by race. J Matern Fetal Med. 2000 Jul-Aug;9(4):238-41. doi: 10.1002/1520-6661(200007/08)9:43.0.CO;2-5. PMID 11048836
- [Background] Woods C. At-risk, pregnant youth and appropriate use of health care. Am Fam Physician. 2010 Mar 1;81(5):577. No abstract available. PMID 20187592